CLINICAL TRIAL: NCT02357654
Title: GnRH for Luteal Support in IVF/ICSI/FET Cycles
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Reproductive Associates (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO20140001128
Record Dates: First submitted 2015-01-07; First posted 2015-02-06 (Estimated); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Gonadotropin-Releasing Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GnRH agonist (Experimental)
  Interventions: Drug: GnRH
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: GnRH — single shot of GnRH agonist
  Arms: GnRH agonist
Drug: placebo — placebo
  Arms: Placebo

SUMMARY:
During IVF cycles an embryo is generally placed into the uterine cavity between 3 and 5 days after fertilization. For a successful pregnancy to take place, that embryo must then implant in the properly primed and staged endometrium, which subsequently must continue to develop to accommodate the growing and maturing embryo and then fetus. This process is normally regulated by hormonal interactions between the fetal, endometrial and luteal tissue. It has been found that after IVF additional support for the endometrium with progesterone improves implantation and subsequent live birth rates in IVF cycle . Recent data has shown that additional supplementation with a single administration of a GnRH agonist around the time the time of embryo transfer may further enhance these rates .

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* women undergoing IVF/ICSI or frozen embryo transfers (FET) that less than 40 years old.

Exclusion Criteria:

* day 3 transfers

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 350 (Estimated)
Dates: Start 2015-11; Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Live birth per transfer | 9 months

SECONDARY OUTCOMES:
implantation rates | 4 weeks
clinical pregnancy | 4 weeks
rates of OHSS | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter G McGovern, MD, Principal Investigator — Rutgers University
Locations (1):
- University Reproductive Associates, Hasbrouck Heights, New Jersey, United States

REFERENCES:
- [Background] van der Linden M, Buckingham K, Farquhar C, Kremer JA, Metwally M. Luteal phase support for assisted reproduction cycles. Cochrane Database Syst Rev. 2011 Oct 5;(10):CD009154. doi: 10.1002/14651858.CD009154.pub2. PMID 21975790
- [Background] Oliveira JB, Baruffi R, Petersen CG, Mauri AL, Cavagna M, Franco JG Jr. Administration of single-dose GnRH agonist in the luteal phase in ICSI cycles: a meta-analysis. Reprod Biol Endocrinol. 2010 Sep 8;8:107. doi: 10.1186/1477-7827-8-107. PMID 20825643

DOCUMENTS (1):
  • Informed Consent Form (2023-10-18): https://cdn.clinicaltrials.gov/large-docs/54/NCT02357654/ICF_000.pdf